CLINICAL TRIAL: NCT01935141
Title: Efficacy Of Low(30 Ml) Versus Full Dose (100 Ml)Contrast CT Pulmonary Angiography Performed On 64 Multi-Detector CT In Detecting Emboli
Brief Title: Efficacy of Low (30ml) Versus Full Dose (100ml) Contrast CT Pulmonary Angiography in Detecting Emboli
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing difficulties to run project.
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bruce Barack, Staff Radiologist, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2012-101526
Record Dates: First submitted 2013-08-21; First posted 2013-09-04 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Pulmonary Emboli
Keywords: Pulmonary Embolus; Radio Contrast Material; Computed Tomography
MeSH Terms: conditions — Pulmonary Embolism | interventions — Contrast Media; iodixanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-Dose IV Contrast (Experimental): A single intravenous dose of 30 ml of Visipaque 320 non-ionic isoosmolar contrast agent will be given for each CT scan. The CT scan will be performed using a Siemens Sensation 64-MDCT scanner.
  Interventions: Procedure: Low-Dose IV Contrast; Device: Siemens Sensation 64-MDCT scanner.; Drug: Visipaque 320 non-ionic isoosmolar contrast agent
- Full-Dose IV Contrast (Active Comparator): A single intravenous dose of 100ml of Visipaque 320 non-ionic isoosmolar contrast agent will be given for each CT scan. The CT scan will be performed using a Siemens Sensation 64-MDCT scanner.
  Interventions: Procedure: Low-Dose IV Contrast; Device: Siemens Sensation 64-MDCT scanner.; Drug: Visipaque 320 non-ionic isoosmolar contrast agent

INTERVENTIONS:
Procedure: Low-Dose IV Contrast — A single intravenous dose of 30 ml of Visipaque (Iodixanol) 320 non-ionic isoosmolar contrast agent will be given for each CT scan.
  Other Names: Visipaque; Iodixanol
Device: Siemens Sensation 64-MDCT scanner. — The device will be used to perform CT Pulmonary Angiograms
Drug: Visipaque 320 non-ionic isoosmolar contrast agent — Single Dose of Intravenous Iodixanol will be administered per CT scan.
  Other Names: Iodixanol

SUMMARY:
With the improvement in CT scanners and injectors, diagnostic chest CT can now be performed in less than 10 seconds. It was hypothesized that diagnostic CT pulmonary angiograms could be done with less than the usual 80-120 ml of contrast used. We have developed a method of performing diagnostic CT pulmonary angiograms with 30 ml of intravenous contrast in most patients. The long-term objective of this study is to show that there is no difference in the diagnostic efficacy of this low dose 30 ml technique when compared to the more traditional full-dose technique.

DETAILED DESCRIPTION:
Potential participants in the study will have been referred to the radiology section for a CTPA for a suspected pulmonary embolus. The radiologist will review the patient's record in CPRS, as is done routinely in this situation. Patients with class 3 or 4 CHF, supraventricular tachycardia, Serum Creatinine >1.5 mg/dl (>1.3 mg/dl female), history of contrast allergy, or unable to give informed consent will be excluded from both arms of the study. Patients with serum creatinine >1.28 mg/dl require referring physician approval. If the participant appears to qualify for the study then the study physician will contact the referring physician and inform him/her of the study. If the referring physician is agreeable then either the radiologist or the referring physician will approach the patient, either at the bedside or in the radiology clinic to determine if the patient is interested in participating in the study. If so, a study radiologist will begin the informed consent process. After informed consent is obtained the subject will be computer randomized to either the new low-dose or full-dose technique protocols. A total of 220 studies (110 per group) will be performed.

Multidetector CT Scan: All CT examinations will be performed on the Siemens Sensation 64-MDCT scanner. Visipaque (Iodixanol) 320 non-ionic isoosmolar contrast agent will be used in all contrast examinations followed by a subsequent injection of normal saline. An informed written consent for the injection of IV contrast will be obtained prior to all CT examinations. Safe venous access will be obtained via either an antecubital vein or a central venous line. For low dose CT pulmonary angiograms, 30 ml of IV Radio Contrast Material (RCM) will be injected at a flow rate of 5 ml/second followed by an injection of 20 ml of normal saline at 5ml/second. The region of interest (ROI) will be the superior vena cava (SVC) at the approximate level of the aortic arch. The scan will be triggered to begin at 75 Hounsfield units (HU). For Full dose CT pulmonary angiograms, 100 ml of IV RCM will be injected at a flow rate of 5ml/sec. The ROI will be the main pulmonary artery. The scan will be triggered at 120 HU. One mm contiguous axial spiral scans will be obtained from the apex of the lung through the adrenals. Reformatted 1.5 mm axial, 3 mm axial, 1.5 mm coronal and sagittal images will be obtained. All images will be uploaded to the AGFA Picture Archiving Communication System (PACS) workstation for interpretation. The costs of all CT scans and RCM will be covered by the Department of Imaging as the majority of the studies are part of routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for CT pulmonary angiogram to exclude pulmonary embolus

Exclusion Criteria:

* Class 3 or 4 Congestive Heart Failure
* Supraventricular tachycardia
* History of contrast allergy
* Unable to give informed consent
* Patients with serum creatinine >1.28 mg/dl without referring physician approval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
CT Image Quality Score | Within 4 weeks of the CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Bruce M. Barack, M.D., Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- VALosAngeles, Los Angeles, California, United States